CLINICAL TRIAL: NCT03324880
Title: A Randomized, Double-blind, Placebo-controlled, Adaptive Study to Evaluate Symptom Improvement and Metabolic Control Among Adult Subjects With Symptomatic Hypoparathyroidism Treated With Recombinant Human Parathyroid Hormone [rhPTH(1-84)]
Brief Title: A Study to Learn if Recombinant Human Parathyroid Hormone [rhPTH(1-84)] Can Improve Symptoms and Metabolic Control in Adults With Hypoparathyroidism (BALANCE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP634-401; 2017-000284-32 (EudraCT Number)
Record Dates: First submitted 2017-10-10; First posted 2017-10-30 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Hypoparathyroidism
Keywords: rhPTH[1-84); Parathyroid hormone; Hypocalcemia; Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to rhPTH (1-84) as subcutaneous (SC) injection once daily (QD) with active vitamin D and calcium supplements up to 31.3 weeks.
  Interventions: Biological: Placebo
- rhPTH (1-84) (Experimental): Participants received rhPTH (1-84) 50 microgram (mcg) SC injection QD, titrated within the dose range of 25-100 mcg QD as an adjunctive treatment with active vitamin D and calcium supplements based on metabolic response up to 32 weeks.
  Interventions: Biological: rhPTH (1-84)

INTERVENTIONS:
Biological: rhPTH (1-84) — rhPTH (1-84) SC injection.
  Arms: rhPTH (1-84)
Biological: Placebo — Placebo QD SC injection.
  Arms: Placebo

SUMMARY:
Recombinant human parathyroid hormone, also known as if rhPTH(1-84), is a medicine to treat people with Hypothyroidism. The main aim of this study is to learn if rhPTH(1-84) can improve symptoms in adults with hypoparathyroidism.

In this study, participants will receive 1 of 2 treatments: rhPTH(1-84) or a placebo. A placebo looks like the medicine being studied but does not have medicine in it. In this study, the placebo will be a standard treatment which is either active Vitamin D, or active Vitamin D with calcium. Active Vitamin D is a form of vitamin D that has a faster effect on the body. These treatments will be given as a daily injection just under the skin. Participants will not know which treatment they received, nor will their study doctors. This is to help make sure the results are more reliable. All participants will also take active vitamin D and calcium supplements during treatment.

Participants will record their symptoms in a tool called the hypoparathyroidism symptom diary. This tool is used to assess symptoms and their impact and will give an overall score for each participant.

The study doctors will also check for side effects from the study treatments.

After treatment, researchers will check if there is any difference in the diary scores between the 2 treatment groups. A difference in score means there is a difference in symptoms and their impact. From this, researchers will learn if symptoms have improved for participants treated with rhPTH(1-84) compared with those treated with placebo.

DETAILED DESCRIPTION:
24 SEPTEMBER 2020: The temporary enrollment stop of new patients into this study due to the COVID-19 pandemic has been lifted in one or more countries, and the study is now again enrolling new patients. However, some countries/sites may still have paused the enrollment of new patients due to the pandemic.

20 APRIL 2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Has an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Is able to voluntarily provide a signed and dated informed consent form before any study-related procedures are performed.
* Is an adult male or female 18 to 85 years of age, inclusive.
* In participants 18-25 years of age, has radiological evidence of epiphyseal closure based on bone age X-ray (single posteroanterior X-ray of left wrist and hand) before randomization.
* Has chronic hypoparathyroidism with onset 12 months or more before screening. The diagnosis of hypoparathyroidism is established based on hypocalcemia in the setting of inappropriately low serum PTH levels.
* During the Week -3 screening visit, the participant reports by history at least 2 of the following symptoms related to hypoparathyroidism occurring within the 2 weeks before Week -3 visit: muscle cramps, muscle spasms or twitching, tingling, numbness, heaviness in arms or legs, physical fatigue, or slowed or confused thinking (brain fog).
* The participant must have a Hypoparathyroidism Symptom Diary (HPT-SD) symptom subscale Sum Score of greater than or equal to (>=) 10 during the 14-day period immediately prior to the baseline (Week 0) visit (Day -14 to Day -1). In addition, the participant must have at least 4 HPT-SD diaries completed in the first 7 day period and at least 4 HPT-SD diaries completed in second 7 day period.
* Must be treated with active vitamin D (calcitriol or alfacalcidol) alone or in conjunction with calcium supplements for at least 4 months prior to the screening visit.

  1. The participant must be taking >= 0.5 microgram (mcg)/day of calcitriol or >=1.0 mcg/day of alfacalcidol.
  2. If the participant is treated with a lower dose of active vitamin D the participant must also be taking calcium supplements of at least 800 milligrams per day (mg/day) of elemental calcium.
* Has serum thyroid-stimulating hormone (TSH) results within normal laboratory limits at screening for all participants not receiving thyroid hormone replacement therapy. For participants on thyroid hormone replacement therapy, the thyroid hormone dose must have been stable for at least 4 weeks before screening, and serum TSH level must be within the central laboratory normal range. A serum TSH level below the lower limit of the normal range but not undetectable in participant treated with thyroid hormone may be allowed if there is no anticipated need for a change in thyroid hormone dose during the trial.
* Has serum 25-hydroxyvitamin D levels >=50 nmol/L (nanomoles per liter) (20 nanograms per milliliter [ng/mL]) and less than (<) 1.5 times the upper limit of normal (ULN) for the central laboratory normal range.
* Has estimated glomerular filtration rate (eGFR) greater than (>) 30 milliliter per minute per 1.73 square meters (ml/min/1.73m^2).
* Prior to randomization, is able to perform daily SC self-injections of study medication (or have a designee perform injection) via a multidose injection pen into the thigh.
* Willing to use oral active vitamin D and calcium supplements provided for the study unless directed to remain on the supplements used prior to enrollment in the current study by the investigator after consultation with the medical monitor.
* With regard to female participants: women who are postmenopausal (12 consecutive months of spontaneous amenorrhea and age >= 51 years) and women who are surgically sterilized can be enrolled. Women of childbearing potential must have a negative pregnancy test at randomization and be willing to comply with any applicable contraceptive requirements of the protocol and pregnancy testing for the duration of the study.

Exclusion Criteria:

* History of hypoparathyroidism resulting from a known activating mutation in the CaSR gene or impaired responsiveness to PTH (pseudohypoparathyroidism).
* Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, such as poorly controlled hyperthyroidism; Paget disease; type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus; severe and chronic cardiac, liver (Child-Pugh score >9) (US FDA, 2003), or renal disease; Cushing syndrome; rheumatoid arthritis; myeloma; active pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy (other than low-risk well differentiated thyroid cancer); primary or secondary hyperparathyroidism; or documented parathyroid carcinoma within the previous 5 years, acromegaly, or multiple endocrine neoplasia types 1 and 2.
* Very low or very high blood calcium level (eg, ACSC <1.87 mmol/L [<7.5 mg/dL] or >=2.97 mmol/L [>=11.9 mg/dL]) at the Week -3 screening visit. Results from the central laboratory must be used for this assessment.
* Blood calcium level above the ULN at the baseline (Week 0) visit. Results from a local laboratory may be used for this assessment.
* Use of prohibited medications, such as loop and thiazide diuretics, phosphate binders (other than calcium carbonate), digoxin, lithium, methotrexate, or systemic corticosteroids, within respective prohibited periods.
* Participation in any other investigational study in which receipt of investigational drug or device occurred within 6 months before screening for this study. Prior treatment with PTH-like drugs (whether commercially available or through participation in an investigational study), including PTH(1-84), PTH(1-34), or other N-terminal fragments or analogs of PTH or PTH-related protein, within 3 months before screening.
* Use of other drugs known to influence calcium and bone metabolism, such as calcitonin, fluoride tablets, or cinacalcet hydrochloride, within the prohibited period.
* Use of oral bisphosphonates within the previous 6 months or intravenous bisphosphonate preparations within the previous 24 months before screening.
* Nonhypocalcemic seizure disorder with a history of a seizure within the previous 6 months before screening. Participants with a history of seizures that occur in the setting of hypocalcemia are allowed.
* The participant is at increased baseline risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, hereditary disorders predisposing to osteosarcoma, or with a prior history of external beam or implant radiation therapy involving the skeleton.
* Any disease or condition that, in the opinion of the investigator, may require treatment or make the participant unlikely to fully complete the study or any condition that presents undue risk from the investigational product or procedures. For example, illness that is anticipated to be chronic and not transient.
* Pregnant or lactating women.
* Known or suspected intolerance or hypersensitivity to the investigational product, closely-related compounds, or any of the stated ingredients.
* History of diagnosed drug or alcohol dependence within the previous 3 years.
* Poorly controlled short bowel syndrome, bowel resection, tropical sprue, celiac disease, ulcerative colitis, and Crohn disease.
* Chronic or severe cardiac disease including but not limited to heart failure (according to the New York Heart Association classification Class II to Class IV) (Dolgin and NYHA, 1994), arrhythmias, bradycardia (resting heart rate <50 beats/minute).
* History of cerebrovascular accident.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (40):
- United States (6):
  - University of Chicago, Chicago, Illinois
  - Michigan Bone and Mineral Clinic, Detroit, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Physicians East PA, Greenville, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Belgium (2):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
- Canada (4):
  - Nova Scotia Health Authority (Capital District Health Authority), Halifax, Nova Scotia
  - Bone Research and Education Centre, Oakville, Ontario
  - CHU de Quebec-Universite Laval, Québec
  - Eastern Health - Health Sciences Center- General Hospital, St. John's
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
  - Odense Universitetshospital, Odense C
- France (4):
  - CHU Angers, Angers
  - Hopital Jean Minjoz, Besançon
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
- Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony, Germany
- Italy (3):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Universita di Firenze, Dipartimento di Chirurgia e Medicina Traslazionale (DCMT), Florence
  - Università Campus Bio Medico Di Roma, Roma
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum, Leiden
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF Rikshospitalet, Oslo
  - Oslo Universitetssykehus Aker, Oslo
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Unidade Local de Saúde de Matosinhos SA, Matosinhos Municipality
  - Centro Hospitalar de São João, E.P.E., Porto
- Spain (4):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- United Kingdom (5):
  - Ninewells Hospital - PPDS, Dundee, Dundee City
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Queen Elizabeth Hospital, Birmingham
  - Leicester Royal Infirmary, Leicester
  - Manchester Royal Infirmary - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Brandi ML, Vokes T, Appelman-Dijkstra NM, Ayodele O, Decallonne B, de Jongh R, Diaz-Curiel M, Fraser W, Finkelman RD, Heck A, Ing SW, Kamenicky P, Khan AA, Kovacs CS, Lapauw B, Leese G, Mantovani G, Martinez Diaz-Guerra G, Masi L, Melo M, Palermo A, Reddy NL, Rejnmark L, Tokareva E, Vantyghem MC, Wang S, Warren M, Yan B. rhPTH(1-84) for hypoparathyroidism: a randomized study of patient-reported outcomes. Eur J Endocrinol. 2025 Jul 31;193(2):310-319. doi: 10.1093/ejendo/lvaf148. PMID 40711996
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fda4db2bf003ab4711e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 35 investigative sites in Belgium, Canada, Denmark, Spain, France, United Kingdom, Italy, Netherlands, Norway, Portugal, Sweden and the United States (US) from 24 January 2018 to 19 May 2022.
Pre-assignment Details: Participants with a diagnosis of symptomatic hypoparathyroidism were enrolled in 1:1 ratio to receive placebo matching rhPTH (1-84) with active vitamin D and/or calcium supplements or rhPTH (1-84) with active vitamin D and/or calcium supplements.
Period: Overall Study
Arm/Group | Placebo | rhPTH (1-84)
Started | 48 | 45
Completed | 46 | 39
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Product Recall | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants in the Intention-to-Treat (ITT) Set who took at least 1 dose of investigational product (study drug or placebo).
Groups:
- Placebo: Participants received placebo matched to rhPTH (1-84) as SC injection QD with active vitamin D and calcium supplements up to 31.3 weeks.
- rhPTH (1-84): Participants received rhPTH (1-84) 50 mcg SC injection QD, titrated within the dose range of 25-100 mcg QD as an adjunctive treatment with active vitamin D and calcium supplements based on metabolic response up to 32 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | rhPTH (1-84) | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.16) | 47.8 (10.41) | 48.5 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 39 | 31 | 70
  Unknown or Not Reported | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 43 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hypoparathyroidism Symptom Diary (HPT-SD/HypoPT-SD) Symptom Subscale Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — HypoPT-SD: 13-item patient-reported outcomes instrument including symptom subscale (items 1-7), anxiety (item 8), sadness/depression (item 9), impact subscale (items 10-13). Items 1-9 score: None=0 to Very severe=4; Items 10-13: Not at all=0 to Very much=2. Item score=average of daily item response over 14-day period before visit. If data were unavailable for at least 4 out of 7 days during both 7-day periods within 14-day period, score was set to missing. Symptom subscale score=average of symptom items 1-7 scores. Symptom subscale score:0 to 4 points with higher scores=more severe symptoms. Population: Number analyzed is the number of participants with data available for analysis.
  score on a scale
    number analyzed (Participants) | 47 | 45 | 92
    (all) | 2.23 (0.541) | 2.56 (0.728) | 2.39 (0.657)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hypoparathyroidism Symptom Diary (HypoPT-SD) Symptom Subscale Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. The symptom subscale score was computed as the average of symptom items 1-7 scores with more than 3 of the 7 symptom item scores were non-missing. Negative change in scores indicates improvement. A mixed model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 26
Population: ITT Set included all randomized participants. Overall number analyzed is the number of participants with data available at the time of analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale | -0.93 (0.130) | -1.46 (0.137)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.003, MMRM — 1-sided p-value was reported; Difference in Least Squares (LS) Mean = -0.53, 95% CI 2-sided [-0.90 to -0.15], Standard Error of Mean 0.189; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD symptom subscale score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD symptom subscale score

2. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 26
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) questionnaire contains 13 fatigue-related questions. The responses to the 13 items on the FACIT-Fatigue questionnaire are each measured on a 5-point Likert scale, where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit and 4=Very much. Thus, the total score ranges from 0 to 52. High scores represent less fatigue. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 28
score on a scale | 4.4 (1.87) | 15.0 (1.93)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 10.5, 95% CI 2-sided [5.1 to 15.9], Standard Error of Mean 2.70; MMRM analysis over all post-baseline visits, with the change from baseline in FACIT-Fatigue total score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline FACIT-Fatigue total score

3. Secondary Outcome: Change From Baseline in Physical Component Summary (PCS) Derived From 36-Item Short Form Health Survey Version 2 (SF-36v2) Scores at Week 26
Description: The SF-36 is a validated instrument that questions participants about perceived physical and mental health and function. The SF-36 consists of 8 scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight; the lower the score the more disability. Change in PCS derived from SF-36v2 at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 29
score on a scale | 4.404 (1.3514) | 8.646 (1.3406)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.015, MMRM — 1-sided p-value was reported; Difference in LS Mean = 4.242, 95% CI 2-sided [0.413 to 8.072], Standard Error of Mean 1.9219; MMRM analysis over all post-baseline visits, with the change from baseline in SF-36 PCS score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline SF-36 PCS score

4. Secondary Outcome: Change From Baseline in Hypoparathyroidism Symptom Diary (HypoPT-SD) Impact Subscale Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. The impact subscale score was computed as the average of impact items 10-13 scores with no impact item score was non-missing. Negative change in scores indicates improvement. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale | -0.36 (0.076) | -0.69 (0.081)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.002, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.32, 95% CI 2-sided [-0.55 to -0.10], Standard Error of Mean 0.112; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD impact subscale score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD impact subscale score

5. Secondary Outcome: Change From Baseline in Individual Hypoparathyroidism Symptom Diary (HypoPT-SD) Impact Items Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. The change in individual symptom item scores was reported. Negative change in scores indicates improvement. MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale
  Impact on Sleep | -0.39 (0.086) | -0.68 (0.090)
  Ability to Exercise | -0.35 (0.088) | -0.71 (0.093)
  Ability to Complete Work | -0.39 (0.084) | -0.76 (0.089)
  Impact Family Relationships | -0.29 (0.083) | -0.66 (0.088)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Impact on Sleep; Test type: Superiority; p = 0.013, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.28, 95% CI 2-sided [-0.53 to -0.04], Standard Error of Mean 0.125; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD impact item score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD impact item score
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Ability to Exercise; Test type: Superiority; p = 0.003, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.36, 95% CI 2-sided [-0.61 to -0.11], Standard Error of Mean 0.128; [other analysis details as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); Ability to Complete Work; Test type: Superiority; p = 0.002, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.36, 95% CI 2-sided [-0.61 to -0.12], Standard Error of Mean 0.123; [other analysis details as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); Impact Family Relationships; Test type: Superiority; p = 0.002, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.37, 95% CI 2-sided [-0.61 to -0.13], Standard Error of Mean 0.121; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Hypoparathyroidism Symptom Diary (HypoPT-SD) Symptom Item Anxiety (Item 8) Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. The anxiety item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the anxiety item score was set to missing. Negative change in scores indicates improvement. MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale | -0.79 (0.139) | -1.35 (0.147)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.004, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.55, 95% CI 2-sided [-0.96 to -0.15], Standard Error of Mean 0.203; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD anxiety item score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD anxiety item score

7. Secondary Outcome: Change From Baseline in Hypoparathyroidism Symptom Diary (HypoPT-SD) Symptom Item Sadness or Depression (Item 9) Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. The sadness or depression item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the item score was set to missing. Negative change in scores indicates improvement. MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale | -0.76 (0.137) | -1.30 (0.145)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.004, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.54, 95% CI 2-sided [-0.93 to -0.14], Standard Error of Mean 0.200; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD sadness or depression item score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD sadness or depression item score

8. Secondary Outcome: Change From Baseline in Individual Hypoparathyroidism Symptom Diary (HypoPT-SD) Symptom Item Scores at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. Negative change in scores indicates improvement. MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 30
score on a scale
  Muscle Cramps | -0.91 (0.150) | -1.47 (0.158)
  Tingling | -1.04 (0.146) | -1.58 (0.154)
  Numbness | -0.89 (0.158) | -1.37 (0.167)
  Muscle Spasms | -0.87 (0.149) | -1.49 (0.159)
  Feelings of Heaviness | -0.96 (0.157) | -1.34 (0.166)
  Physical Fatigue | -0.89 (0.155) | -1.45 (0.165)
  Brain Fog | -0.90 (0.127) | -1.40 (0.134)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Muscle Cramps; Test type: Superiority; p = 0.006, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.56, 95% CI 2-sided [-0.99 to -0.12], Standard Error of Mean 0.218; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD symptom item score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD symptom item score
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Tingling; Test type: Superiority; p = 0.007, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.54, 95% CI 2-sided [-0.96 to -0.12], Standard Error of Mean 0.213; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.020, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.48, 95% CI 2-sided [-0.94 to -0.02], Standard Error of Mean 0.231; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); Muscle Spasms; Test type: Superiority; p = 0.003, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.62, 95% CI 2-sided [-1.05 to -0.18], Standard Error of Mean 0.219; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs rhPTH (1-84); Feelings of Heaviness; Test type: Superiority; p = 0.050, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.38, 95% CI 2-sided [-0.83 to 0.07], Standard Error of Mean 0.229; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs rhPTH (1-84); Physical Fatigue; Test type: Superiority; p = 0.008, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.55, 95% CI 2-sided [-1.01 to -0.10], Standard Error of Mean 0.227; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs rhPTH (1-84); Brain Fog; Test type: Superiority; p = 0.004, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.51, 95% CI 2-sided [-0.87 to -0.14], Standard Error of Mean 0.186; [other analysis details as in outcome 8, analysis 1]

9. Secondary Outcome: Number of Participants With Response at Week 26 [Early Termination (ET)]
Description: Response was defined as a 30% reduction in HypoPT-SD symptom subscale score from baseline. The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4; and for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. The symptom subscale score was computed as the average of symptom items 1-7 scores with more than 3 of the 7 symptom item scores were non-missing. Data reported also includes results for early terminated participants.
Time Frame: Baseline up to Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 32
Participants | 24 | 25

10. Secondary Outcome: Change From Baseline in the Most Bothersome Symptom Score at Week 26
Description: The HypoPT-SD is a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness or depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None=0 to Very severe=4 and for items 10-13, it ranges from Not at all=0 to Very much=2. An item score was computed by taking the average of the daily item response over the 14-day period immediately before the visit. If data were not available for at least 4 out of 7 days during both 7-day periods within the 14-day period, the individual item score was set to missing. The Most Bothersome Symptom Score was analyzed. Negative change in scores indicates improvement. MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 38 | 26
score on a scale | -0.87 (0.156) | -1.77 (0.174)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.90, 95% CI 2-sided [-1.37 to -0.43], Standard Error of Mean 0.235; MMRM analysis over all post-baseline visits, with the change from baseline in HypoPT-SD most bothersome symptom score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect, with adjustment for baseline HypoPT-SD most bothersome symptom score

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) Perceived Cognitive Impairments (PCI) Score at Week 26
Description: The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) assessment is a 37-item instrument. The perceived cognitive impairment and the impact on quality of life domains were assessed in this study. These 2 domains include 22 items rated on a 5-point scale. The perceived cognitive impairments subscale contains 18 items and each item has a 5-point ordinal response scale (0=Never, 1= About once a week, 2 = Two to three times a week, 3= Nearly every day, 4 = Several times a day). Each item score is calculated as (4 minus item response), and the subscale score is [sum of (4 minus item response)]*18/(number of items answered)]. The perceived cognitive impairment subscale score ranges from 0 to 72, with higher scores indicate better cognitive function. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 28
score on a scale | 2.7 (0.74) | 4.8 (0.76)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.024, MMRM — 1-sided p-value was reported; Difference in LS Mean = 2.1, 95% CI 2-sided [0.0 to 4.3], Standard Error of Mean 1.07; MMRM analysis over all post-baseline visits, with the change from baseline in FACT-Cog Perceived Cognitive Impairments Subscale score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline FACT-Cog Perceived Cognitive Impairments Subscale score

12. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) Impact on Quality of Life (QoL) Score at Week 26
Description: The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) assessment is a 37-item instrument. The perceived cognitive impairment and the impact on quality of life domains were assessed in this study. These 2 domains include 22 items rated on a 5-point scale. The impact on quality of life domain contains 4 items and each item has a 5-point ordinal response scale (0=Never, 1= About once a week, 2 = Two to three times a week, 3= Nearly every day, 4 = Several times a day). Each item score is calculated as (4 minus item response), and the subscale score is [sum of (4 minus item response)]*4/(number of items answered)]. The impact on quality of life subscale score ranges from 0 to 16 with higher score indicates better cognitive function. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 28
score on a scale | 2.7 (0.74) | 4.8 (0.76)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.024, MMRM — 1-sided p-value was reported; Difference in LS Mean = 2.1, 95% CI 2-sided [0.0 to 4.3], Standard Error of Mean 1.07; MMRM analysis over all post-baseline visits, with the change from baseline in FACT-Cog QoL Subscale score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline FACT-Cog QoL Subscale score

13. Secondary Outcome: Change From Baseline in Individual Domains of 36-Item Short Form Health Survey Version 2 (SF-36v2) at Week 26
Description: The SF-36 is a validated instruments that question participants about perceived physical and mental health and function. The SF-36 consists of 8 scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight; the lower the score the more disability. Change in the score of individual domains of SF-36v2 at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: ITT Set included all randomized participants. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available analysis for specified categories.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 29
score on a scale
  Standard-Bodily Pain | 4.194 (1.4987) | 11.404 (1.4919)
  Standard-General Health | 3.515 (1.4509) | 9.061 (1.4463)
  Standard-Mental Health | 3.719 (1.6098) | 11.576 (1.6043)
  Standard-Physical Functioning | 4.833 (1.4850) | 9.387 (1.4669)
  Standard-Role-Emotional | 5.228 (1.6322) | 13.648 (1.6254)
  Standard-Role-Physical | 5.964 (1.5799) | 10.194 (1.5670)
  Standard-Social Functioning | 6.005 (1.8636) | 9.814 (1.8661)
  Standard-Vitality | 4.205 (1.6539) | 12.147 (1.6547)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Standard-Bodily Pain; Test type: Superiority; p = 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 7.210, 95% CI 2-sided [2.951 to 11.469], Standard Error of Mean 2.1376; MMRM analysis over all post-baseline visits, with the change from baseline in SF-36 domain score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline SF-36 domain score
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Standard-General Health; Test type: Superiority; p = 0.004, MMRM — 1-sided p-value was reported; Difference in LS Mean = 5.545, 95% CI 2-sided [1.452 to 9.638], Standard Error of Mean 2.0542; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); Standard-Mental Health; Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 7.857, 95% CI 2-sided [3.292 to 12.423], Standard Error of Mean 2.2913; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); Standard-Physical Functioning; Test type: Superiority; p = 0.017, MMRM — 1-sided p-value was reported; MMRM = 4.554, 95% CI 2-sided [0.345 to 8.763], Standard Error of Mean 2.1123; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs rhPTH (1-84); Standard-Role-Emotional; Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 8.420, 95% CI 2-sided [3.800 to 13.040], Standard Error of Mean 2.3186; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs rhPTH (1-84); Standard-Role-Physical; Test type: Superiority; p = 0.032, MMRM — 1-sided p-value was reported; Difference in LS Mean = 4.230, 95% CI 2-sided [-0.251 to 8.711], Standard Error of Mean 2.2489; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs rhPTH (1-84); Standard-Social Functioning; Test type: Superiority; p = 0.079, MMRM — 1-sided p-value was reported; Difference in LS Mean = 3.809, 95% CI 2-sided [-1.502 to 9.121], Standard Error of Mean 2.6658; [other analysis details as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs rhPTH (1-84); Standard-Vitality; Test type: Superiority; p = 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 7.942, 95% CI 2-sided [3.253 to 12.630], Standard Error of Mean 2.3530; [other analysis details as in outcome 13, analysis 1]

14. Secondary Outcome: Change From Baseline in Mental Component Summary (MCS) Score of 36-Item Short Form Health Survey Version 2 (SF-36v2) at Week 26
Description: The SF-36 is a validated instruments that question participants about perceived physical and mental health and function. The SF-36 consists of 8 scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight; the lower the score the more disability. Change in the MCS of SF-36v2 at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 29
score on a scale | 4.297 (1.5898) | 12.597 (1.5904)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value; Difference in LS Mean = 8.300, 95% CI 2-sided [3.788 to 12.811], Standard Error of Mean 2.2642; MMRM analysis over all post-baseline visits, with the change from baseline in SF-36 MCS score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline SF-36 MCS score

15. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Hypoparathyroidism (WPAI: Hypoparathyroidism) Score at Week 26
Description: WPAI assessed impact of HypoPT on work productivity and daily activities. Concepts that WPAI: Hypoparathyroidism measures include time missed from work and impairment of work and other regular activities due to specific health problem (HypoPT). WPI was calculated based on 4 items including Q2: hours of work missed due to HPT; Q4: actual hours worked; Q5: HPT effect on productivity at work; Q6: HPT effect on daily activities. Scores for 4 subscales were calculated as Percent work time missed due to problem: Q2/(Q2+Q4)*100; Percent impairment while working due to problem: Q5/10*100; Percent overall work impairment due to problem: Q2/(Q2+Q4)+[(1(Q2/(Q2+Q4)))x(Q5/10)]*100; Percent activity impairment due to problem: Q6/10*100. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. Change from baseline in questionnaire response was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: ITT Set included all randomized participants. Overall number analyzed is the number of participants with data available at the time of analyses. Number analyzed is the number of participants with data available for analysis for specified categories.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 29 | 27
score on a scale
  Percent Work Time Missed Due to Problem: number analyzed (Participants) | 15 | 11
  Percent Work Time Missed Due to Problem | 2.30 (6.279) | 5.43 (7.155)
  Percent Impairment While Working Due to Problem: number analyzed (Participants) | 14 | 9
  Percent Impairment While Working Due to Problem | -11.7 (4.79) | -26.3 (5.76)
  Percent Overall Work Impairment Due to Problem: number analyzed (Participants) | 14 | 9
  Percent Overall Work Impairment Due to Problem | -11.17 (3.854) | -26.08 (4.774)
  Percent Activity Impairment Due to Problem | -10.2 (3.97) | -23.3 (4.17)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Percent Work Time Missed Due to Problem; Test type: Superiority; p = 0.627, MMRM — 1-sided p-value was reported; Difference in LS Mean = 3.13, 95% CI 2-sided [-16.33 to 22.60], Standard Error of Mean 9.578; MMRM analysis over all post-baseline visits, with the change from baseline in WPAI score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline WPAI score
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Percent Impairment While Working Due to Problem; Test type: Superiority; p = 0.031, MMRM — 1-sided p-value was reported; Difference in LS Mean = -14.6, 95% CI 2-sided [-29.9 to 0.7], Standard Error of Mean 7.52; [other analysis details as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); Percent Overall Work Impairment Due to Problem; Test type: Superiority; p = 0.011, MMRM — 1-sided p-value was reported; Difference in LS Mean = -14.90, 95% CI 2-sided [-27.42 to -2.39], Standard Error of Mean 6.146; [other analysis details as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); Percent Activity Impairment Due to Problem; Test type: Superiority; p = 0.014, MMRM — 1-sided p-value was reported; Difference in LS Mean = -13.0, 95% CI 2-sided [-24.5 to -1.5], Standard Error of Mean 5.78; [other analysis details as in outcome 15, analysis 1]

16. Secondary Outcome: Change From Baseline in Scores of Patient's Assessment of Overall Health Status Using Patient Global Impression of Severity (PGI-S) at Week 26
Description: The PGI-S is a global index that can be used to rate the severity of a specific condition. The PGI-S is a rating scale that asks the respondent to best describe how their symptoms severity. Response options are assessed as per 5-point scale: no symptoms (0), mild (1), moderate (2), severe (3), and very severe (4). Mean change in scores of PGI-S at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 34 | 29
score on a scale | -0.8 (0.15) | -1.4 (0.16)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.010, MMRM — 1-sided p-value; Difference in LS Mean = -0.5, 95% CI 2-sided [-1.0 to -0.1], Standard Error of Mean 0.22; MMRM analysis over all post-baseline visits, with the change from baseline in PGI-S score as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline PGI-S score

17. Secondary Outcome: Change From Baseline in Scores of Patient's Assessment of Overall Health Status Using Patient Global Impression of Change (PGI-C) at Week 26
Description: The PGI-C is verbal rating scale asks the respondent to best describe change in symptoms compared to the beginning of study. Response options are assessed using a 7-point scale: very much improved (0), much improved (1), minimally improved (2), no change (3), minimally worse (4), much worse (5), and very much worse (6). Negative change indicates improvement. Mean change in scores of PGI-C at Week 26 was be reported.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 30 | 28
score on a scale | -0.6 (1.04) | -1.7 (1.63)

18. Secondary Outcome: Change From Baseline in In-Clinic Neurocognitive Assessment Scores at Week 24
Description: Neurocognitive test battery included tests evaluating frontal-executive domain, which encompasses functions attributable to prefrontal cortex and its connections to basal ganglia (mostly striatum). Tests included the CogState (CS) Brief Battery (including the Detection: speed [range from 2.001 to 6; lower scores (LS) indicate improvement (IMP)], Identification: speed [range from 2.001 to 6; LS indicate IMP], One Card Learning: accuracy [range from 0 to 1.5708; higher scores (HS) indicate IMP], One Back: speed [range from 2.001 to 6; LS indicate IMP]), CS Groton Maze Learning Test: total errors (range from 0 to infinity; LS indicate IMP), CS International Shopping List Task (ISLT): number of correct responses (range from 0 to infinity; HS indicate IMP), and CS ISLT -Delayed Recall: number of correct responses (range from 0 to infinity; HS indicate IMP). Change in in-clinic neurocognitive assessment scores at Week 24 was reported. Analysis of Covariance (ANCOVA) was used for analysis.
Time Frame: Baseline, Week 24
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 34 | 30
score on a scale
  Detection | 0.03 [0.01 to 0.06] | 0.05 [0.02 to 0.08]
  Identification: number analyzed (Participants) | 33 | 30
  Identification | 0.02 [-0.01 to 0.05] | 0.04 [0.01 to 0.07]
  One Card Learning: number analyzed (Participants) | 33 | 30
  One Card Learning | 0.12 [0.07 to 0.16] | 0.13 [0.08 to 0.17]
  One Back (ONB): number analyzed (Participants) | 33 | 30
  One Back (ONB) | 0.09 [0.06 to 0.12] | 0.09 [0.06 to 0.13]
  Groton Maze Learning (GML): number analyzed (Participants) | 33 | 30
  Groton Maze Learning (GML) | -2.43 [-9.89 to 5.02] | 7.49 [-0.46 to 15.45]
  International Shopping List (ISL) | 1.98 [0.73 to 3.24] | 1.42 [0.08 to 2.76]
  International Shopping List Test Delayed Recall (ISRL): number analyzed (Participants) | 32 | 28
  International Shopping List Test Delayed Recall (ISRL) | 1.31 [0.62 to 1.99] | 1.86 [1.13 to 2.59]
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Detection; Test type: Superiority; p = 0.516, ANCOVA; From an Analysis of Covariance (ANCOVA) with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.03 to 0.05]
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Identification; Test type: Superiority; p = 0.275, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 0.02, 95% CI 2-sided [-0.02 to 0.06]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); One Card Learning; Test type: Superiority; p = 0.777, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.05 to 0.07]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); One Back (ONB); Test type: Superiority; p = 0.831, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.04 to 0.05]
Statistical Analysis 5: Comparison: Placebo vs rhPTH (1-84); Groton Maze Learning (GML); Test type: Superiority; p = 0.075, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 9.93, 95% CI 2-sided [-1.00 to 20.85]
Statistical Analysis 6: Comparison: Placebo vs rhPTH (1-84); International Shopping List (ISL); Test type: Superiority; p = 0.545, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = -0.57, 95% CI 2-sided [-2.41 to 1.27]
Statistical Analysis 7: Comparison: Placebo vs rhPTH (1-84); International Shopping List Test Delayed Recall (ISRL); Test type: Superiority; p = 0.283, ANCOVA; From an ANCOVA with treatment group (rhPTH(l-84), placebo) as the predictor and Baseline score as a covariate; Difference in LS Mean = 0.55, 95% CI 2-sided [-0.45 to 1.56]

19. Secondary Outcome: Change From Baseline in At-Home Neurocognitive Assessment Scores at Week 26
Description: Neurocognitive test battery included tests evaluating frontal-executive domain, which encompasses functions attributable to prefrontal cortex and its connections to basal ganglia (mostly striatum). Tests included the CogState (CS) Brief Battery (including the Detection: speed [range from 2.001 to 6; lower scores (LS) indicate improvement (IMP)], Identification: speed [range from 2.001 to 6; LS indicate IMP], One Card Learning: accuracy [range from 0 to 1.5708; higher scores (HS) indicate IMP], One Back: speed [range from 2.001 to 6; LS indicate IMP]). Changes in at-home neurocognitive assessment scores (CS Brief Battery) at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 45 | 38
score on a scale
  Detection (DET): number analyzed (Participants) | 45 | 37
  Detection (DET) | -0.01 [-0.03 to 0.00] | -0.01 [-0.03 to 0.01]
  Identification (IDN) | -0.01 [-0.03 to 0.01] | 0.00 [-0.02 to 0.02]
  One Card Learning (OCL): number analyzed (Participants) | 45 | 37
  One Card Learning (OCL) | 0.08 [0.05 to 0.11] | 0.09 [0.06 to 0.12]
  One Back (ONB) | 0.02 [0.00 to 0.04] | 0.03 [0.01 to 0.05]
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Detection (DET); Test type: Superiority; p = 0.582, MMRM — 1-sided p-value was reported; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.02 to 0.04]; From MMRM with visit, treatment group, and visit treatment group as fixed effects, Baseline score as a covariate, and participant as a random effect. By-participant scores, which are summarized in this table, are derived as the average of the planned at-home assessment values that passed the Completion criteria over 14 days preceding the visit
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Identification (IDN); Test type: Superiority; p = 0.492, MMRM — 1-sided p-value was reported; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.02 to 0.04]; [other analysis details as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs rhPTH (1-84); One Card Learning (OCL); Test type: Superiority; p = 0.506, MMRM — 1-sided p-value was reported; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.03 to 0.06]; [other analysis details as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs rhPTH (1-84); One Back Test; Test type: Superiority; p = 0.438, MMRM — 1-sided p-value was reported; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.02 to 0.04]; [other analysis details as in outcome 19, analysis 1]

20. Secondary Outcome: Change From Baseline in 24-hour Urine Calcium Excretion at Week 26
Description: Change in 24-hour urine calcium excretion at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per day (mmol/day)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 43 | 33
millimoles per day (mmol/day) | -1.99 (0.574) | 0.11 (0.651)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.991, MMRM — 1-sided p-value was reported; Difference in LS Mean = 2.09, 95% CI 2-sided [0.36 to 3.83], Standard Error of Mean 0.871; MMRM analysis over all post-baseline visits, with the change from baseline in 24-hour urine calcium excretion as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline 24-Hour urine calcium excretion

21. Secondary Outcome: Change From Baseline in Serum Phosphate Level at Week 26
Description: Change in serum phosphate level at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 47 | 40
millimoles per liter (mmol/L) | 0.030 (0.0270) | -0.145 (0.0289)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = -0.175, 95% CI 2-sided [-0.254 to -0.097], Standard Error of Mean 0.0395; MMRM analysis over all post-baseline visits, with the change from baseline in serum phosphate as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline serum phosphate

22. Secondary Outcome: Change From Baseline in Doses of Active Vitamin D at Week 26
Description: Changes in doses of active vitamin D at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: micrograms per day (μg/day)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 47 | 38
micrograms per day (μg/day) | -5.65 (3.155) | -1.57 (3.418)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.810, MMRM — 1-sided p-value was reported; Difference in LS Mean = 4.08, 95% CI 2-sided [-5.06 to 13.22], Standard Error of Mean 4.654; From a mixed-effects model for repeated measures (MMRM) analysis over all post-baseline visits, with the change from baseline in active vitamin D supplement dose as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline active vitamin D supplement dose

23. Secondary Outcome: Change From Baseline in Doses of Calcium Supplements at Week 26
Description: Changes in doses of calcium supplements at Week 26 was reported. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per day (mg/day)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 47 | 40
milligrams per day (mg/day) | -44.3 (91.13) | -375.6 (96.20)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p = 0.007, MMRM — 1-sided p-value was reported; Difference in LS Mean = -331.3, 95% CI 2-sided [-594.6 to -67.9], Standard Error of Mean 132.56; MMRM analysis over all post-baseline visits, with the change from baseline in elemental calcium supplement dose as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline elemental calcium supplement dose

24. Secondary Outcome: Change From Baseline in Albumin-corrected Serum Calcium Control at Week 26
Description: Change From Baseline in albumin-corrected serum calcium between 1.875 millimoles per liter (mmol/L) (7.5 milligram per deciliter [mg/dL]) and upper limit of normal (ULN) for the central laboratory normal range at Week 26 was reported.
Time Frame: Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 47 | 40
mmol/L | -0.033 (0.2072) | 0.090 (0.2254)

25. Secondary Outcome: Number of Participants Who Achieve Composite Criteria for Albumin-corrected Serum Calcium Concentration, Active Vitamin D Dose and Oral Elemental Calcium Supplement Dose at Week 26
Description: Number of participants achieving composite criteria of the following: albumin-corrected serum calcium between 1.875 mmol/L (7.5 mg/dL) and the ULN for the central laboratory normal range, dose of active vitamin D decreased by 50% and at least a 50% reduction from the baseline oral elemental calcium supplement dose at Week 26 was reported.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 47 | 40
Participants | 6 | 21

26. Secondary Outcome: Change From Baseline in Bone Turnover Marker Bone Specific Alkaline Phosphatase at Week 26
Description: Bone turnover markers included serum bone-specific alkaline phosphatase, procollagen amino-terminal peptide, C-terminal telopeptide of type 1 collagen, and osteocalcin. A MMRM was used for analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units per liter (U/L)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 44 | 37
units per liter (U/L) | 0.69 (2.256) | 23.03 (2.365)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 22.33, 95% CI 2-sided [15.83 to 28.84], Standard Error of Mean 3.271; MMRM analysis over all post-baseline visits, with the change from baseline in bone turnover biomarkers as the outcome, treatment group, visit, and their interaction as fixed effect factors and participants as a random effect with adjustment for baseline bone turnover biomarkers

27. Secondary Outcome: Change From Baseline in Bone Turnover Marker Type I Collagen C-Telopeptides at Week 26
Description: as for outcome 26
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanograms per liter (ng/L)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 45 | 36
nanograms per liter (ng/L) | -5.0 (76.52) | 780.5 (84.00)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 785.5, 95% CI 2-sided [559.6 to 1011.3], Standard Error of Mean 113.65; [other analysis details as in outcome 26, analysis 1]

28. Secondary Outcome: Change From Baseline in Bone Turnover Marker Osteocalcin and Procollagen 1 N-Terminal Propeptide at Week 26
Description: as for outcome 26
Time Frame: Baseline, Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: micrograms per liter (µg/L)
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 45 | 36
micrograms per liter (µg/L)
  Osteocalcin | -0.88 (4.109) | 55.55 (4.476)
  Procollagen 1 N-Terminal Propeptide: number analyzed (Participants) | 45 | 34
  Procollagen 1 N-Terminal Propeptide | 1.95 (22.744) | 228.52 (24.475)
Statistical Analysis 1: Comparison: Placebo vs rhPTH (1-84); Osteocalcin; Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 56.43, 95% CI 2-sided [44.33 to 68.53], Standard Error of Mean 6.091; [other analysis details as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs rhPTH (1-84); Procollagen 1 N-Terminal Propeptide; Test type: Superiority; p < 0.001, MMRM — 1-sided p-value was reported; Difference in LS Mean = 226.57, 95% CI 2-sided [160.17 to 292.98], Standard Error of Mean 33.425; [other analysis details as in outcome 26, analysis 1]

29. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as AEs that started or worsened on or after the date and time of the first dose of investigational product.
Time Frame: From start of study drug administration to 4 weeks post follow-up (up to Week 36)
Population: Safety Analysis Set included all participants in the ITT Set who took at least 1 dose of investigational product (study drug or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | rhPTH (1-84)
Number analyzed (Participants) | 48 | 45
Participants | 46 | 41

ADVERSE EVENTS:
Time Frame: From start of study drug administration to 4 weeks post follow-up (up to Week 36)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included all participants in the ITT Set who took at least 1 dose of investigational product (study drug or placebo).
Arm/Group | Placebo | rhPTH (1-84)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 6/48 | 6/45
Other Adverse Events (participants affected / at risk) | 41/48 | 38/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | rhPTH (1-84) (N=45)
Anxiety (Psychiatric disorders) | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3
Sinusitis (Infections and infestations) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | rhPTH (1-84) (N=45)
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Depression (Psychiatric disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Dizziness (Nervous system disorders) | 6 | 5
Fatigue (General disorders) | 4 | 5
Feeling abnormal (General disorders) | 1 | 5
Gastroenteritis (Infections and infestations) | 2 | 3
Headache (Nervous system disorders) | 11 | 14
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 4
Hypertension (Vascular disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Influenza (Infections and infestations) | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Nasopharyngitis (Infections and infestations) | 7 | 4
Nausea (Gastrointestinal disorders) | 9 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Palpitations (Cardiac disorders) | 5 | 1
Paraesthesia (Nervous system disorders) | 5 | 6
Urinary tract infection (Infections and infestations) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03324880/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03324880/SAP_001.pdf